CLINICAL TRIAL: NCT01849835
Title: A Test of the Comparison Between Trans-rectal and Trans-perineal Biopsy of Prostate
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Le-hang Guo, Principal Investigator, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: tongji10us; tongji10-us1
Record Dates: First submitted 2013-04-29; First posted 2013-05-09 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Complication
Keywords: rate of positive detection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trans-rectal (Experimental): trans-rectal to perform the prostate biopsy
  Interventions: Procedure: trans-rectal to perform the prostate biopsy
- trans-perineal (Experimental): trans-perineal to perform the prostate biopsy
  Interventions: Procedure: trans-perineal to perform the prostate biopsy

INTERVENTIONS:
Procedure: trans-rectal to perform the prostate biopsy — the puncture points are at the rectal
  Arms: trans-rectal
Procedure: trans-perineal to perform the prostate biopsy — the puncture points are at the perineal
  Other Names: the puncture points are at the perineal
  Arms: trans-perineal

SUMMARY:
The purpose of this randomized controlled trial (RCT) is to compare the two ways (tras-rectal and trans-perineal) to perform prostate biopsy from the rate of Positive detection, complications, pain level, operation time and costs et al.

ELIGIBILITY:
Inclusion Criteria:

* prostate-specific antigen > 4ng/ml
* Palpation is positive

Exclusion Criteria:

* older than 80y
* prostate-specific antigen > 100 ng/ml

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
the rate of positive detections | 1year

SECONDARY OUTCOMES:
the incidence rate of each complication | 1 year

OTHER OUTCOMES:
pain level assessed by visual analogue scale | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- 10Th Hospital of Tongji University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Evidence-based Guidelines for Best Practice in Health Care Transrectal Ultrasound Guided Biopsy of the Prostate